CLINICAL TRIAL: NCT00876694
Title: A 52-week Treatment, Multi-center, Randomized, Open Label, Parallel Group Study to Assess the Long Term Safety and Efficacy of Indacaterol (300 µg o.d.) Using Salmeterol (50 µg b.i.d.) as an Active Control in Japanese Patients With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Confirmatory Study of Indacaterol in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CQAB149B1303
Record Dates: First submitted 2009-04-03; First posted 2009-04-07 (Estimated); Results first posted 2011-11-08 (Estimated); Last update posted 2011-11-08 (Estimated); Status verified 2011-10

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: COPD, Chronic Obstructive Pulmonary Disease, Indacaterol, long acting β2-agonist
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — indacaterol; Salmeterol Xinafoate

ARMS (2):
- Indacaterol 300 µg (Experimental): Indacaterol 300 μg once a day (o.d.) delivered via single dose dry powder inhaler (SDDPI). Daily ICS monotherapy, if needed, was allowed to remain stable throughout study. Salbutamol was available for rescue use throughout study.
  Interventions: Drug: Indacaterol 300 µg
- Salmeterol 50 µg (Active Comparator): Salmeterol 50 μg twice a day (b.i.d.) delivered via Diskus®. Daily ICS monotherapy, if needed, was allowed to remain stable throughout study. Salbutamol was available for rescue use throughout study.
  Interventions: Drug: Salmeterol 50 µg

INTERVENTIONS:
Drug: Indacaterol 300 µg — Indacaterol 300 µg once daily (od) via SDDPI
  Arms: Indacaterol 300 µg
Drug: Salmeterol 50 µg — Salmeterol 50 µg twice daily (bid) via Diskus®
  Arms: Salmeterol 50 µg

SUMMARY:
This study is designed to collect long term safety data of indacaterol (300 µg o.d.) in Japanese patients with moderate to severe COPD. Data from this study will be used for the registration of indacaterol in Japan.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of COPD (moderate-to-severe as classified by the Global Initiative for Chronic Obstructive Lung Disease (GOLD) Guidelines) and:

* Smoking history of at least 20 pack-years
* Post-bronchodilator FEV1 <80% and ≥30% of the predicted normal value
* Post-bronchodilator FEV1/FVC (forced vital capacity) <70%

Exclusion Criteria:

1. Patients who have been hospitalized for a COPD exacerbation in the 6 weeks prior to Visit 1 or during the run-in period
2. Patients who have had a respiratory tract infection within 6 weeks prior to Visit 1
3. Patients with concomitant pulmonary disease
4. Patients with a history of asthma
5. Patients with diabetes Type I or uncontrolled diabetes Type II
6. Any patient with lung cancer or a history of lung cancer
7. Patients with a history of certain cardiovascular comorbid conditions
8. Patients who have been exposed to indacaterol previously. (Except for any patient who enrolled in Study CQAB149B1302)

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Actual)
Dates: Start 2009-03; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (37):
- Japan (37):
  - Novartis Investigator Site, Asahikawa
  - Novartis Investigator Site, Bunkyō City
  - Novartis Investigator Site, Gifu
  - Novartis Investigator Site, Hamamatsu
  - Novartis Investigator Site, Himeji
  - Novartis Investigator Site, Hiroshima
  - Novartis Investigator Site, Iwata
  - Novartis Investigator Site, Kanazawa
  - Novartis Investigator Site, Kasaoka
  - Novartis Investigator Site, Kawasaki
  - Novartis Investigator Site, Kishiwada
  - Novartis Investigator Site, Kitakyushu
  - Novartis Investigator Site, Kochi
  - Novartis Investigator Site, Koga
  - Novartis Investigator Site, Kurume
  - Novartis Investigator Site, Kyoto
  - Novartis Investigator Site, Maebashi
  - Novartis Investigator Site, Matsusaka
  - Novartis Investigator Site, Morioka
  - Novartis Investigator Site, Nagaoka
  - Novartis Investigator Site, Nagoya
  - Novartis Investigator Site, Naka-gun
  - Novartis Investigator Site, Noda
  - Novartis Investigator Site, Obihiro
  - Novartis Investigator Site, Sakai
  - Novartis Investigator site, Sapporo
  - Novartis Investigator Site, Sendai
  - Novartis Investigator Site, Setagaya-ku
  - Novartis Investigator Site, Sumida-ku
  - Novartis Investigator Site, Tenri
  - Novartis Investigator Site, Tokyo
  - Novartis Investigator Site, Ube
  - Novartis Investigator Site, Wakayama
  - Novartis Investigator Site, Yabu
  - Novartis Investigator Site, Yanagawa
  - Novartis Investigator Site, Yokkaichi
  - Novartis Investigator Site, Yokohama

RESULTS

PARTICIPANT FLOW:
Groups:
- Indacaterol 300 μg: Indacaterol 300 μg once a day (o.d.) delivered via single dose dry powder inhaler (SDDPI). Daily ICS monotherapy, if needed, was allowed to remain stable throughout study. Salbutamol was available for rescue use throughout study.
- Salmeterol 50 μg: Salmeterol 50 μg twice a day (b.i.d.) delivered via Diskus®. Daily ICS monotherapy, if needed, was allowed to remain stable throughout study. Salbutamol was available for rescue use throughout study.
Period: Overall Study
Arm/Group | Indacaterol 300 μg | Salmeterol 50 μg
Started | 125 | 61
Completed | 104 | 49
Not Completed | 21 | 12
Not completed — Adverse Event | 10 | 7
Not completed — Subject withdrew consent | 6 | 4
Not completed — Unsatisfactory therapeutic effect | 2 | 0
Not completed — Abnormal test procedure result(s) | 1 | 0
Not completed — Administrative problems | 1 | 1
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Indacaterol 300 μg | Salmeterol 50 μg | Total
Number analyzed (Participants) | 125 | 61 | 186
Age Continuous [Mean (Standard Deviation); unit: years] | 70 (7.81) | 67.3 (8.05) | 69.1 (7.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 1 | 10
  Male | 116 | 60 | 176

OUTCOME MEASURES:

1. Primary Outcome: The Number of Participants With a Clinically Notable Pulse Rate During 52 Weeks of Treatment
Description: The number of participants with newly occurring or worsening clinically notable vital sign: Pulse Rate in beats per minute (bpm) at anytime post baseline (BL) by treatment. Low Pulse Rate was defined as a pulse rate <40 bpm or <= to 50 bpm and a decrease from baseline >= to 15 bpm. High Pulse Rate was defined as a pulse rate >130 bpm or >= to 120 bpm and an increase from baseline >= to 15 bpm.
Time Frame: 52 weeks
Population: The safety population included all patients who received at least one dose of study drug.
Measure: Number; unit: Participants
Arm/Group | Indacaterol 300 μg | Salmeterol 50 μg
Number analyzed (Participants) | 125 | 61
Participants
  Low Pulse Rate: | 1 | 0
  High Pulse Rate: | 0 | 0

2. Primary Outcome: The Number of Participants With a Clinically Notable Systolic Blood Pressure During 52 Weeks of Treatment
Description: The number of participants with newly occurring or worsening clinically notable vital sign: Systolic Blood Pressure (mmHg) at anytime post baseline (BL) by treatment.
  A Low Systolic Blood Pressure was defined as a systolic blood pressure measurement: <75 mmHg or <= to 90 mmHg and a decrease from baseline >= to 20 mmHg.
  A High Systolic Blood Pressure was defined as a systolic blood pressure measurement: >200 mmHg or >= to 180 mmHg and an increase from baseline >= to 20 mmHg.
Time Frame: 52 weeks
Population: The safety population included all patients who received at least one dose of study drug.
Measure: Number; unit: Participants
Arm/Group | Indacaterol 300 μg | Salmeterol 50 μg
Number analyzed (Participants) | 125 | 61
Participants
  Low Systolic Blood Pressure: | 0 | 0
  High Systolic Blood Pressure: | 1 | 0

3. Primary Outcome: The Number of Participants With a Clinically Notable Diastolic Blood Pressure During 52 Weeks of Treatment
Description: The number of participants with newly occurring or worsening clinically notable vital sign: Diastolic blood pressure (mmHg) at anytime post baseline (BL) by treatment.
  A Low Diastolic Blood Pressure was defined as a diastolic blood pressure measurement: <40 mmHg or <= to 50 mmHg and a decrease from baseline >= to 15 mmHg.
  A High Diastolic Blood Pressure was defined as a diastolic blood pressure measurement: >115 mmHg or >= to 105 mmHg and an increase from baseline >= to 15 mmHg.
Time Frame: 52 weeks
Population: The safety population included all patients who received at least one dose of study drug.
Measure: Number; unit: Participants
Arm/Group | Indacaterol 300 μg | Salmeterol 50 μg
Number analyzed (Participants) | 125 | 61
Participants
  Low Diastolic Blood Pressure: | 0 | 1
  High Diastolic Blood Pressure: | 0 | 0

4. Primary Outcome: The Number of Participants With a Clinically Notable QTc Interval Value During 52 Weeks of Treatment
Description: The number of participants with newly occurring or worsening clinically notable QTc Interval value at anytime post baseline.
  The QTc interval is calculated using Fridericia's formula: QTc= QT/cube root RR. QTc is the interval between the Q and T waves corrected for heart rate and RR is the interval between two R waves in milliseconds (ms).
  Notable QTc interval >450 ms for males and >470 ms for females. The maximum QTc increase from baseline at any time during the study was also tabulated with absolute and relative frequencies for categories 30- 60 ms and >60 ms.
Time Frame: 52 weeks
Population: The safety population included all patients who received at least one dose of study drug.
Measure: Number; unit: Participants
Arm/Group | Indacaterol 300 μg | Salmeterol 50 μg
Number analyzed (Participants) | 125 | 61
Participants
  Notable QTc | 6 | 3
  QTc increase from BL: 30-60 ms | 12 | 3
  QTc increase from BL: >60 ms | 0 | 1

5. Primary Outcome: Serum Potassium (mmol/L) at Weeks 4, 8, 12, 24, 36, 44, and 52
Description: The least squares mean of the serum potassium in mmol/L at weeks 4, 8, 12, 24, 36, 44 and 52. Mixed model used baseline serum potassium as a covariate.
Time Frame: 4, 8, 12, 24, 36, 44, and 52 weeks
Population: The safety population included all patients who received at least one dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Indacaterol 300 μg | Salmeterol 50 μg
Number analyzed (Participants) | 125 | 61
mmol/L
  Week 4 (n= 122, 57) | 4.26 (0.028) | 4.28 (0.039)
  Week 8 (n= 121, 56) | 4.30 (0.032) | 4.27 (0.044)
  Week 12 (n= 118, 56) | 4.28 (0.033) | 4.35 (0.044)
  Week 24 (n= 113, 52) | 4.34 (0.035) | 4.27 (0.048)
  Week 36 (n= 106, 50) | 4.35 (0.032) | 4.29 (0.044)
  Week 44 (n= 104, 50) | 4.31 (0.033) | 4.27 (0.044)
  Week 52 (n= 104, 49) | 4.32 (0.035) | 4.31 (0.048)

6. Primary Outcome: Blood Glucose (mmol/L) 1 Hour Post Dose at Weeks 4, 8, 12, 24, 36, 44, and 52
Description: The least squares mean of the blood glucose in mmol/L at weeks 4, 8, 12, 24, 36, 44 and 52. Mixed model used baseline blood glucose as a covariate.
Time Frame: 4, 8, 12, 24, 36, 44, and 52 weeks
Population: The safety population included all patients who received at least one dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Indacaterol 300 μg | Salmeterol 50 μg
Number analyzed (Participants) | 125 | 61
mmol/L
  Week 4 (n= 122, 57) | 6.10 (0.187) | 5.96 (0.260)
  Week 8 (n= 121, 56) | 5.92 (0.159) | 6.30 (0.220)
  Week 12 (n= 118, 56) | 5.97 (0.199) | 6.59 (0.262)
  Week 24 (n= 113, 52) | 6.16 (0.195) | 6.13 (0.271)
  Week 36 (n= 106, 50) | 5.95 (0.137) | 6.26 (0.189)
  Week 44 (n= 104, 50) | 6.09 (0.226) | 6.42 (0.309)
  Week 52 (n= 104, 49) | 5.96 (0.220) | 6.65 (0.296)

7. Secondary Outcome: Trough Forced Expiratory Volume in 1 Second (FEV1) After 12, 24 and 52 Weeks
Description: Trough FEV1 was defined as the mean of the values at 23 h 10 min and 23 h 45 min after dosing at clinic on the previous day. Trough FEV1 was analyzed after 12, 24 and 52 weeks using a mixed model which contained the baseline FEV1 measurement, FEV1 prior to inhalation and FEV1 30 minutes post inhalation of salbutamol as covariates.
Time Frame: After 12, 24 and 52 weeks
Population: The intention-to-treat (ITT) population included all randomized patients who received at least one dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Indacaterol 300 μg | Salmeterol 50 μg
Number analyzed (Participants) | 125 | 61
Liters
  Week 12 (n= 122, 56) | 1.40 (0.013) | 1.33 (0.019)
  Week 24 (n= 112, 51) | 1.40 (0.016) | 1.34 (0.022)
  Week 52 (n= 105, 49) | 1.39 (0.017) | 1.31 (0.023)

ADVERSE EVENTS:
Time Frame: 52 weeks
Description: Safety population.
Arm/Group | Indacaterol 300 μg | Salmeterol 50 μg
Serious Adverse Events (participants affected / at risk) | 16/125 | 4/61
Other Adverse Events (participants affected / at risk) | 61/125 | 26/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Indacaterol 300 μg (N=125) | Salmeterol 50 μg (N=61)
Angina pectoris (Cardiac disorders) | 1 | 0
Retinal haemorrhage (Eye disorders) | 0 | 1
Uveitis (Eye disorders) | 0 | 1
Colonic polyp (Gastrointestinal disorders) | 1 | 0
Sudden death (General disorders) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 3 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Meniscus lesion (Injury, poisoning and procedural complications) | 1 | 0
Computerised tomogram abnormal (Investigations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebral infarction (Nervous system disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Arteriosclerosis obliterans (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Indacaterol 300 μg (N=125) | Salmeterol 50 μg (N=61)
Bronchitis (Infections and infestations) | 5 | 4
Nasopharyngitis (Infections and infestations) | 34 | 13
Upper respiratory tract infection (Infections and infestations) | 8 | 3
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 26 | 14
Cough (Respiratory, thoracic and mediastinal disorders) | 14 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.